CLINICAL TRIAL: NCT00437749
Title: Phase 3, Randomized, Double-Blind, Placebo-controlled Study of CBT-1 and Paclitaxel/Carboplatin in Patients With Inoperable Non-Small Cell Lung Cancer
Brief Title: A Study of CBT-1 and Paclitaxel With Carboplatin in Patients With Advanced Inoperable Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow accrual rate; interim accrual objective met
Sponsor: CBA Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBA-TP0301
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non small cell lung cancer; Advanced; Inoperable; taxanes; carboplatin; multi-drug resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- CBT-1 (Active Comparator)
  Interventions: Drug: CBT-1
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBT-1 — (50 mg caps) 500 mg/m2/day x 7 + paclitaxel 135 mg/m2 + carboplatin AUC 6
  Arms: CBT-1
Other: Placebo — (50 mg caps) 500 mg/m2/day x 7 + paclitaxel 135 mg/m2 + carboplatin AUC 6
  Arms: Placebo

SUMMARY:
Multiple Drug Resistance is the phenomena whereby cells become resistant to a variety of drugs with different mechanisms of action. Drug resistance remains a significant impediment to successful cancer chemotherapy inhibitors have been developed and are currently in clinical trials. CBT-1 is a natural product currently in clinical trials as an inhibitor

DETAILED DESCRIPTION:
Lung cancer has the highest incidence and prevalence among cancers in the world and remains the leading cause of cancer-related deaths in Western countries. One-year survival of patients with best supportive care remains low. Non-small-cell lung cancer accounts for almost 85% of all lung cancer cases. Approximately 70% of patients have locally advanced or metastatic disease at presentation and are not candidates for surgery.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed diagnosis of NSCLC
* advanced inoperable NSCLC
* have adequate renal function, serum creatinine <2.0 mg/dL or 24 hour creatinine clearance > 50mL/minute
* have adequate liver function defined as SGOT <4 times the upper limit of normal (ULN) and bilirubin <2.0 mg/dL
* have calcium <11.0 mg/dL and albumin >2.0g/dL
* have adequate bone marrow reserve defined as granulocyte count >1,500/mm3, hemoglobin >10.0 g/dL and platelets >100,000/mm3
* if female and of child-bearing potential, agree to use one of the following methods of birth control: oral contraceptives, barrier with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection, complete abstinence from sexual intercourse

Exclusion Criteria:

* have previously received taxanes, platinums, vinca alkaloids, anthracyclines, epipodophyllotoxins or CBT-1
* have known or suspected hypersensitivity to platinum containing compounds, taxanes, polyoxyethylated castor oil, or mannitol
* have significant central nervous system disease, including history of seizures within last 3 months or psychiatric history which would impair the ability to give informed consent or prevent compliance with protocol requirements
* be eligible for curative surgery or radiotherapy.
* must not have a diagnosis and/or treatment in the past 5 years of any malignancy other than NSCLC or basal cell carcinoma of the skin
* be pregnant or nursing
* have a history of significant coronary artery disease, cardiac arrhythmias requiring treatment, history of other cardiac disease or other cardiac anomalies determined by ECG which in the judgment of the investigator would compromise the patient's ability to tolerate the therapy
* have ongoing serious infections that require parenteral antibiotics
* have clinically significant bleeding disorders
* have solid organ allograft
* have significant intercurrent disease
* have bleeding peptic ulcer disease
* have participated in any experimental study within 2 months preceding enrollment
* be using a medication that could interact adversely with CBT-1, paclitaxel, or carboplatin. Medications include:aminoglycoside antibiotics, Prilosec, Losec, Zantac

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2001-08; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall Survival | every month for first 6 months off study, then every 2-3 months for the next year, then every 6 months thereafter

SECONDARY OUTCOMES:
Time to Progression | each month for the first 6 months off study, then every 2-3 months for the next year, then every 6 months thereafter.
Response Rates | every 2-3 months following completion of therapy until disease progression
Progression Free Survival | every month for first 6 months off study, then every 2-3 months for next year, then every 6 months thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Oldham, MD, Principal Investigator — CBA Research
Locations (1):
- Arizona Clinical Research Center, Tuscon, Arizona, United States